CLINICAL TRIAL: NCT07001176
Title: Effect of Acute Caffeine Intake on Muscle and Cerebral Oxygenation During Muscular Strength, Power, and Endurance Performance
Brief Title: Caffeine, Resistance Exercise and Muscle/Cerebral Oxygenation
Acronym: CAF+RE+Oxy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CEID/2023/3/070
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Caffeine and Resistance Exercise
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): Acute caffeine intake (3 mg/kg)
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): Acute placebo intake
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — Acute caffeine intake (3 mg/kg)
  Arms: Caffeine
Dietary Supplement: Placebo — Acute placebo intake (3 mg/kg)
  Arms: Placebo

SUMMARY:
Introduction: Several studies have evaluated and confirmed the ergogenic effects of acute caffeine intake on sports performance. However, the mechanism responsible for this ergogenic effect remains to be elucidated.

Objectives: This study aims to evaluate the acute effects of caffeine intake on muscle and cerebral oxygen during muscular strength, power, muscle endurance performance. and muscle electrical activity in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years.
* Body Mass Index (BMI) < 25 kg/m².
* Resistance-trained individuals (more than 2 years of structured training).
* Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from exercising.
* Participants must be able to perform the tests described in the following section.

Exclusion Criteria:

* History of neuromuscular diseases, heart disease, or conditions that may affect liver or muscle metabolism.
* Use of drugs, stimulants, or sports supplements that could interfere with the dietary supplement used in the study.
* Sedentary habits (less than 150 minutes/week of moderate exercise).
* Having undergone prolonged periods of physical inactivity in the 6 months prior to the study.
* Engaging in strenuous exercise within 48 hours prior to the tests.
* Failure to replicate the same food intake on both experimental days.
* Consumption of caffeine or any other stimulant after 6 pm on the day before the tests, to avoid headaches, discomfort, or lethargy in regular caffeine consumers.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Muscle Oxygenation | Through study completion, an average of 2 weeks
  Measuring oxygen in the muscle before and after exercise.
Cerebral oxygenation | Through study completion, an average of 2 weeks
  Measuring cerebral oxygenation before and after exercise.
Number of repetitions performed in 1 set at 65%1RM until task failure | Through study completion, an average of 2 weeks
Bar velocity deplacement performed in 1 set at 65%1RM until task failure | Through study completion, an average of 2 weeks
  In bench press and back squat exercises
Power output generated in 1 set at 65%1RM until task failure | Through study completion, an average of 2 weeks
  In bench press and back squat exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes